CLINICAL TRIAL: NCT06495697
Title: Plasma Pharmacological Monitoring of M Penicillins in Methicillin-sensitive Staphylococcus Aureus Bacteremia - Single-center Retrospective Study
Brief Title: Plasma Pharmacological Monitoring of M Penicillins in Methicillin-sensitive Staphylococcus Aureus Bacteremia
Acronym: DOSESACLOXA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9023
Record Dates: First submitted 2024-04-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-04

CONDITIONS: Staphylococcus Aureus Infection
Keywords: Staphylococcus aureus Infection; Staphylococcus aureus bacteremia; Penicillins; Methicillin-sensitive; Cefazolin; Infectious endocarditis; Staphylococcal endocarditis; Oxacillin; Nephrotoxicity
MeSH Terms: conditions — Staphylococcal Infections; Endocarditis, Subacute Bacterial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The treatment of Methicillin-sensitive Staphylococcus aureus bacteremia is based on the first-line use of cefazolin or M penicillins (oxacillin and cloxacillin). The use of the latter is recommended at high doses (150-200 mg/kg/24h). In a study on infectious endocarditis, 52 of 56 patients with staphylococcal endocarditis treated with (cl)oxacillin were overdosed with the recommended doses. Although the main mechanism of renal toxicity described for M penicillins is immunoallergic, a frequent overdose is observed in cases of acute renal failure with M penicillins. There is also a significant association between overdose and risk of neurological toxicity. The currently recommended treatment duration is a minimum of 14 days of IV treatment from the first negative blood culture, which leaves room for carrying out a plasma assay and possible dosage adjustment subsequently.

Overdose is a risk factor for nephrotoxicity and neurotoxicity. Plasma level could be predictive of clinical success. Systematic plasma dosing would reduce the risk of toxicity and improve the clinical cure rate.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old)
* Having presented an infection with Staphylococcus aureus and treated at the University Hospitals of Strasbourg between January 1, 2019 and December 31, 2022.

Exclusion Criteria:

- Patient having expressed his opposition to the reuse of his data for scientific research purposes.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patient (≥18 years old) having presented an infection with Staphylococcus aureus and treated at the University Hospitals of Strasbourg between January 1, 2019 and December 31, 2022.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-07-19 (Estimated)

PRIMARY OUTCOMES:
Clinical healing | day 30 after infection
  Blood culture negative at 48-96 hours compared to the start of antibiotic therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales - CHU de Strasbourg - France, Strasbourg, France